CLINICAL TRIAL: NCT00462332
Title: Phase II Pilot Trial to Evaluate the Efficacy of a Combined Therapy Approach for Young CLL Patients With Advanced and Progressive Disease Stratified According to the Biological Prognostic Features
Brief Title: Fludarabine and Alemtuzumab or Cyclophosphamide Followed by Peripheral Blood Stem Cell Transplant or Alemtuzumab in Treating Patients With Advanced or Progressive Chronic Lymphocytic Leukemia
Acronym: LLC0405
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LLC0405; LLC0405 (Other: GIMEMA); 2005-002476-15 (EudraCT Number)
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-08

CONDITIONS: Leukemia
Keywords: stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; Alemtuzumab; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High risk patientes (Experimental): Category of risk will be defined according to biological features.
  Interventions: Drug: Fludarabine; Drug: Campath; Procedure: Transplant
- Low risk patients (Experimental): Category of risk will be defined according to biological features.
  Interventions: Drug: Fludarabine; Drug: Campath

INTERVENTIONS:
Drug: Fludarabine — Induction therapy
  Arms: High risk patientes
Drug: Campath — Induction therapy
  Arms: High risk patientes
Procedure: Transplant — Post-induction therapy
  Arms: High risk patientes
Drug: Campath — Post-induction therapy
  Arms: High risk patientes
Drug: Fludarabine — Induction therapy
  Arms: Low risk patients
Drug: Campath — Induction therapy
  Arms: Low risk patients
Drug: Campath — Post-induction therapy
  Arms: Low risk patients

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. A peripheral stem cell transplant using stem cells from the patient or a donor may replace the patient's immune cells that were destroyed by chemotherapy.

PURPOSE: This phase II trial is studying how well giving fludarabine together with alemtuzumab or cyclophosphamide followed by peripheral blood stem cell transplant or alemtuzumab works in treating patients with advanced or progressive chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of induction therapy comprising fludarabine phosphate with either alemtuzumab or cyclophosphamide followed by peripheral blood stem cell transplantation or alemtuzumab in patients with advanced or progressive chronic lymphocytic leukemia.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the length of survival, event-free survival, and disease-free survival of patients treated with this regimen.
* Evaluate the relationship between different clinical and biological disease characteristics, therapeutic response, and survival.

OUTLINE: This is a pilot, multicenter study. Patients are stratified according to biological risk profile (high vs low risk).

* Group 1 (high-risk patients):

  * Induction therapy: Patients receive fludarabine phosphate IV and alemtuzumab IV on days 1-3. Treatment repeats for 4 courses.

Patients with no response (no good clinical partial response, steady disease, or progressive disease) after induction therapy are removed from the study. Other patients proceed to post-induction therapy based on response to induction therapy.

* Post-induction therapy:

  * Complete clinical, cytometric, and molecular response: Patients undergo peripheral blood stem cell (PBSC) mobilization with cytarabine IV twice daily on days 1-3 and filgrastim (G-CSF) followed by no further therapy.
  * Response to induction therapy and evidence of residual disease (complete clinical and cytometric response with molecular evidence of disease; complete clinical response only; or good clinical partial response): Patients without an HLA familial matched donor undergo PBSC mobilization with cytarabine IV twice daily on days 1-3 and G-CSF. Patients with sufficient harvested autologous PBSCs undergo autologous PBSC transplantation (with BEAM conditioning regimen [carmustine, etoposide, cytarabine, and melphalan]). Patients without sufficient harvested
  * PBSCs receive alemtuzumab subcutaneously (SC) weekly for 6 weeks. Patients who do not achieve molecular remission after 6 weeks of alemtuzumab receive 6 additional weeks of treatment. Patients with an HLA familial matched
  * undergo reduced-intensity allogeneic stem cell transplantation (with cyclophosphamide, thiotepa, and fludarabine phosphate as conditioning regimen).

    * Group 2 (low-risk patients):
* Induction therapy: Patients receive fludarabine phosphate and cyclophosphamide on days 1-3. Treatment repeats every month for 4 courses. Patients achieving at least a partial response receive 2 additional courses.

Patients achieving complete clinical response with cytometric and molecular response; complete clinical response with a cytometric response; or complete clinical response after completion of induction therapy (i.e., partial response or greater) receive no further treatment. Patients with no response or disease progression proceed to post-induction therapy.

* Post-induction therapy: Patients receive alemtuzumab SC weekly for 6 weeks. Patients who do not achieve complete remission after 6 weeks of alemtuzumab receive 6 additional weeks of treatment.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia (CLL)

  * Advanced or progressive disease with ≥ 2 active clinical signs

PATIENT CHARACTERISTICS:

* Fertile patients must use adequate contraception
* No positive Coomb's test with signs of hemolysis
* No active infection
* No uncontrolled severe disease
* No known hypersensitivity or anaphylactic reactions to murine antibodies or proteins
* No other malignancies within the past 2 years except for adequately treated malignancies
* No significant traumatic injury within the past 4 weeks
* No coexisting medical or psychological condition that would limit study compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior treatment for CLL
* No major surgery within the past 4 weeks
* No prior chemotherapy

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2007-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Foa, MD, Principal Investigator — Universita Degli Studi "La Sapeinza"
Locations (23):
- Italy (23):
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Universita Degli Studi di Bari, Bari
  - Universita Cattolica del Sacro Cuore - Campobasso, Campobasso
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Ospedale Regionale A. Pugliese, Catanzaro
  - Ospedale Civile Cosenza, Cosenza
  - Universita di Ferrara, Ferrara
  - Azienda Ospedaliera di Firenze, Florence
  - Ospedale San Martino, Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Azienda Ospedaliera Papardo, Messina
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera - Universitaria di Modena, Modena
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome
  - Ospedale Sant' Eugenio, Rome
  - Università Degli Studi "La Sapienza", Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - Azienda Sanitaria Ospedale San Giovanni Battista Molinette di Torino, Turin
  - Policlinico Universitario Udine, Udine

REFERENCES:
- See also: GIMEMA Foundation Website — http://www.gimema.it

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Risk Patientes | Low Risk Patients
Started | 45 | 41
Completed | 45 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Risk Patientes | Low Risk Patients | Total
Number analyzed (Participants) | 45 | 41 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 41 | 86
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 53.02 (6.09) | 52.73 (6.24) | 53.02 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 34 | 28 | 62
Region of Enrollment [Number; unit: participants]
  Italy | 45 | 41 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Response
Description: * Normal clinical or X-ray examination (lymph nodes, liver, spleen)
  * No symptoms
  * Lymphocytes higher or equal to 4.0 per 10^9/L
  * Neutrophils lower or equal to 1.5 per 10^9/L
  * Platelets >100 per 10^9/L
  * Hb >11.0 g/dL
  * Bone marrow lymphs according to age, lymphocytes <30%, no nodules.
Time Frame: At 2 years from study entry
Measure: Number; unit: participants
Arm/Group | Low Risk Patients | High Risk Patients
Number analyzed (Participants) | 41 | 45
participants | 14 | 3

2. Secondary Outcome: Toxicity
Description: Number of AEs and SAEs
Time Frame: At 2 years from study entry
Reporting Status: Not Posted

3. Secondary Outcome: Length of Survival
Time Frame: At 2 years and a half from study entry
Measure: Mean (Standard Deviation); unit: years
Arm/Group | High Risk Patientes | Low Risk Patients
Number analyzed (Participants) | 45 | 41
years | 1.57 (10) | 1.1 (10)

4. Secondary Outcome: Event-free Survival
Time Frame: At 2 years from study entry
Reporting Status: Not Posted

5. Secondary Outcome: Disease-free Survival
Time Frame: At 2 years from study entry
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | High Risk Patientes | Low Risk Patients
Serious Adverse Events (participants affected / at risk) | 7/45 | 9/41
Other Adverse Events (participants affected / at risk) | 32/45 | 33/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Risk Patientes (N=45) | Low Risk Patients (N=41)
Grade >=3 hematologic toxicity (Blood and lymphatic system disorders) | 7 (8) | 9 (10)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Risk Patientes (N=45) | Low Risk Patients (N=41)
AEs related to Campath infusion (Blood and lymphatic system disorders) | 13 (77) | 0 (0)
Infections (Blood and lymphatic system disorders) | 13 (33) | 12 (20)
Hematologic Toxicity (Grade >=3) (Blood and lymphatic system disorders) | 18 (39) | 25 (71)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No